CLINICAL TRIAL: NCT06802445
Title: The Effect of Non-Invasive Vagal Nerve Stimulation Combined With Self-Managed Therapy in Individuals With Myogenic Temporomandibular Dysfunction: A Double-Blind, Randomised, Placebo-Controlled, Clinical Study
Brief Title: The Effect of Non-Invasive Vagal Nerve Stimulation Combined With Self-Managed Therapy in Individuals With Myogenic Temporomandibular Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toros University (Other)
Responsible Party: Principal Investigator, Ümit YÜZBAŞIOĞLU, Lecturer, Toros University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TU-FTR-UY-01
Record Dates: First submitted 2025-01-19; First posted 2025-01-31 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Temporomandibular Disorders (TMD)
Keywords: myogenic temporomandibular disorders; transcutaneous vagal nerve stimulation; pain; self-menaged therapy; posture; muscle activation; muscle stiffness
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain

STUDY DESIGN:
Intervention Model Description: "A Double-Blind, Randomised, Placebo-Controlled, Clinical Study"
  Within the scope of this single-centre, prospective, double-blind, parallel group, placebo-controlled study design, participants will be randomised to 3 groups via a web-based randomisation website.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-Management Therapy Group (Active Comparator): The self-administered therapy programme will consist of prevention of parafunctional activities, information about sleep hygiene and home exercise programmes, the effectiveness of which has been reported in the literature and is in line with the International Delphi Guidelines. Home exercises will start with 2 times a day, 8 repetitions and progress will be made weekly according to the patient's condition.
  Interventions: Other: Self-Management Therapy
- Self-Managed Therapy + Placebo Non-Invasive Vagal Nerve Stimulation (Placebo Comparator): For Placebo Non-Invasive Auricular Transcutaneous Vagal Nerve Stimulation, the technique will be similar to active stimulation. The VaguStim device will be set to 0 Hz by the practitioner, indicating that no actual stimulation is being delivered. Patients will be told that they will not be able to feel the current due to its lower intensity during the intervention, without explaining the true nature of the placebo stimulation.
  Interventions: Other: Self-Management Therapy; Device: Placebo Non-Invasive Vagal Nerve Stimulation
- Self-Managed Therapy + Non-Invasive Vagal Nerve Stimulation (Experimental): Non-Invasive Auricular Transcutaneous Vagal Nerve Stimulation, CE certified (CE No: 2460) non-invasive stimulation device will be applied with. The application will be performed with 3 different sized electrodes (small, medium, large) specially designed according to the size of the inner ear. The stimulation will be delivered bilaterally from the symba concha and tragus regions innervated by the auricular branch of the n.vagus, which guarantees effective and targeted vagal modulation. With reference to the studies in the literature; VaguStim application frequency will be 25 Hz, pulse width 250 µs, current level 0.5 mA with biphasic waveform.
  The treatment will continue 3 days a week for a total of 6 weeks, with each session lasting 20 minutes.
  Interventions: Other: Self-Management Therapy; Device: Non-Invasive Vagal Nerve Stimulation

INTERVENTIONS:
Other: Self-Management Therapy — Participants in this group will receive self management therapy. The self-administered therapy programme will consist of prevention of parafunctional activities, information about sleep hygiene and home exercise programmes, the effectiveness of which has been reported in the literature and is in line with the International Delphi Guidelines. Home exercises will start with 2 times a day, 8 repetitions and progress will be made weekly according to the patient's condition.
Device: Placebo Non-Invasive Vagal Nerve Stimulation — Participants in this group will receive self managemenet therapy and placebo vagal nerve stimulation. For Placebo Non-Invasive Auricular Transcutaneous Vagal Nerve Stimulation, the technique will be similar to active stimulation. The VaguStim device will be set to 0 Hz by the practitioner, indicating that no actual stimulation is being delivered. Patients will be told that they will not be able to feel the current due to its lower intensity during the intervention, without explaining the true nature of the placebo stimulation.
  Arms: Self-Managed Therapy + Placebo Non-Invasive Vagal Nerve Stimulation
Device: Non-Invasive Vagal Nerve Stimulation — Participants will receive Non-Invasive Vagal Nerve Stimulation and self management therapy. : Non-Invasive Auricular Transcutaneous Vagal Nerve Stimulation, CE certified (CE No: 2460) non-invasive stimulation device will be applied with. The application will be performed with 3 different sized electrodes (small, medium, large) specially designed according to the size of the inner ear. The stimulation will be delivered bilaterally from the symba concha and tragus regions innervated by the auricular branch of the n.vagus, which guarantees effective and targeted vagal modulation. With reference to the studies in the literature; VaguStim application frequency will be 25 Hz, pulse width 250 µs, current level 0.5 mA with biphasic waveform. The treatment will continue 3 days a week for a total of 6 weeks, with each session lasting 20 minutes.
  Arms: Self-Managed Therapy + Non-Invasive Vagal Nerve Stimulation

SUMMARY:
The aim of our study is to determine the benefit of non-invasive Vagal Nerve Stimulation in combination with self-administered therapy on the symptoms associated with jaw joint dysfunction in individuals with jaw joint dysfunction.

If you agree to participate in the study, you will fill out a form containing your information such as age, height, body weight. Then, Visual Analog Scale (VAS) and Central Sensitisation Scale will be used to assess the severity of jaw and neck joint pain. The 8-question Jaw Function Restriction Scale will be used to assess the limitation of jaw function.

An algometer will be used to evaluate the pressure-pain threshold, and Therabite range of motion scale will be used to evaluate the range of motion of the jaw joint. One photograph will be taken from the side profile to evaluate the head-neck posture, this photograph will be used for craniocervical angle measurement and will not be shared elsewhere. Myotonmetry will be used to evaluate muscle mechanical properties and non-invasive superficial electromyography (yEMG) will be used to evaluate muscle activation.

The treatments to be applied within the scope of the study will be carried out 3 days a week and the evaluation sessions will last 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-45,
* Diagnosed with myogenic TMDs according to TMD-DC Axis I and II criteria,
* Pain intensity of 3 or more during rest and/or chewing according to the Visual Analogue Scale,
* Volunteered to participate in the study and signed the informed consent form,
* Individuals who do not have communication difficulties and whose native language is Turkish will be included in the study.

Exclusion Criteria:

* Diagnosed with arthrogenic or mixed type TMDs,
* Severe psychiatric illness such as schizophrenia,
* Previous vagal nerve stimulation or history of vagotomy,
* Have extensive joint damage affecting the jaw, head, neck and shoulder areas, have a history of major trauma, fracture or surgery to these body parts, or are undergoing radiotherapy,
* Diagnosed with cervical disc herniation, cervical radiculopathy or cervical myelopathy,
* History of cardiac disease and being treated for cardiac problems,
* Active implant users such as pacemakers, defibrillators, neurostimulators, cochlear implants and ventricular shunts,
* Failure to understand the study protocol
* Have a history of progressive neurological diseases (such as Parkinson's disease, MS, ALS, epilepsy, Alzheimer's disease)
* Acute tinnitus
* Skin problems such as dermatitis, infection, psoriasis, urticaria, acne or eczema at the stimulation site,
* Has any anatomical abnormality that prevents successful placement of the ear electrode,
* and reporting acute tinnitus,
* Pregnant subjects will be excluded from the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-02-08 (Actual); Primary Completion 2026-01-22 (Estimated); Study Completion 2026-02-03 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | First Interview: Initial Assessment/ End of Week 2: Second Evaluation /End of Week 6: Third Evaluation /At the end of Week 12: Fourth and final assessment
  Jaw and neck joint pain intensity will be assessed using the Visual Analogue Scale (VAS),which is reported to be valid and reliable.The individuals included in the study will be asked to indicate the jaw and neck joint pain intensity they have experienced at rest and during chewing in the last 1 week on a 100 mm long line positioned vertically.The marked points will be measured and recorded in millimetres.An increase in VAS indicates pain of higher intensity Pressure-pain threshold measurement will be performed using a digital algometer.Before starting the tests, the individuals will be informed about the test and one trial session will be performed. The tests will be performed using a 1 cm2 headgear with a 1 kg/cm2 increase in pressure intensity every second and the participants will be asked to tell the evaluator the point at which the pressure to be applied turns into mild pain. The average of three consecutive tests performed at 30 s intervals will be taken and recorded in kg/cm2.

SECONDARY OUTCOMES:
Evaluation of Temporomandibular Joint Range of Motion | First Interview: Initial Assessment/ End of Week 2: Second Evaluation /End of Week 6: Third Evaluation /At the end of Week 12: Fourth and final assessment
  The TheraBite® Range of Motion Scale (TheraBite ®, Platon Medikal Ltd., United Kingdom) will be used to assess the range of motion of the participants' jaw joint. TheraBite is a scale with high intra-observer reliability that is frequently used in the literature for the assessment of jaw joint range of motion and is accepted as the standard for clinical use. Participants will be placed supine on a therapy table in an examination room and asked to open their mouths as far as they can and the range of motion will be recorded in millimetres (mm). The measurements will be repeated three times and the average of the three measurements will be taken as reference.Higher values obtained from this scale represent an increase in the range of motion of the mouth.
Craniocervical Posture Assessment | First Interview: Initial Assessment/ End of Week 2: Second Evaluation /End of Week 6: Third Evaluation /At the end of Week 12: Fourth and final assessment
  The craniocervical postures of the individuals included in the study will be evaluated using photogrammetry method based on angle calculation on photographs. For the measurement, the seventh cervical vertebral processes and ear tragus of the individuals will be determined as reference points and these points will be clearly marked before photographing. After the marking is completed, the individual will be asked to perform neck flexion and extension repeatedly to ensure neutral head position in the standing position, and then photographed with a mobile phone camera placed on a tripod 1.5 metres away from the left side of the individual. A craniocervical angle of less than 50 degrees means a forward head posture.
Muscle Activity Measurements | First Interview: Initial Assessment/ End of Week 2: Second Evaluation /End of Week 6: Third Evaluation /At the end of Week 12: Fourth and final assessment
  In the study, a 4-channel superficial EMG (yEMG) device (Ultium EMG Sensor, Noraxon, USA), which is reported to be valid and reliable, will be used to evaluate the activation of masticatory muscles (masseter and temporalis).
Muscle Stiffness | First Interview: Initial Assessment/ End of Week 2: Second Evaluation /End of Week 6: Third Evaluation /At the end of Week 12: Fourth and final assessment
  Stiffness [N/m], is a biomechanical property of a muscle, provides information about the resistance of the tissue to an external force or contraction. stiffness will be measured using a myotonometer (MyotonPRO, Myoton AS, Tallinn, Estonia), which has been reported to be valid and reliable. Assessments will be conducted in study, masseter, upper trapezius, tibialis anterior muscles.The measurement will be repeated 3 times and the arithmetic mean of the measurements will be recorded.
Logarithmic Decrease | First Interview: Initial Assessment/ End of Week 2: Second Evaluation /End of Week 6: Third Evaluation /At the end of Week 12: Fourth and final assessment
  Logarithmic decrease (D) gives information about the elasticity of the evaluated tissue. Logarithmic decrease will be measured using a myotonometer (MyotonPRO, Myoton AS, Tallinn, Estonia), which has been reported to be valid and reliable.Assessments will be conducted in study, masseter, upper trapezius, tibialis anterior muscles.The measurement will be repeated 3 times and the arithmetic mean of the measurements will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Aydan AYTAR, PhD, Study Chair — University of Health Sciences (Ankara-Turkey)
Locations (1):
- Toros University 45 Evler Campus, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No